CLINICAL TRIAL: NCT02813031
Title: Nutritional Intervention Study to Evaluate the Effect of an Olive Oil Lipid Rich in Diglycerides as a Fat Replacement in Different Meat Products, in a Healthy Population
Brief Title: Human Study of Functional Meat Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Principal Investigator, Viviana Loria Kohen, Senior Researcher, Nutrition PhD in Medicine, IMDEA Food
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMD PI014
Record Dates: First submitted 2016-06-17; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: functional meat products; hypocaloric fats; diglyceride; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Functional meat products with healthy lipids from olive oil (Experimental): Healthy people consuming 300g/week of functional meat products with high diglyceride lipid from olive oil
  Interventions: Other: Functional meat products
- Traditional meat products (Placebo Comparator): Healthy people consuming the same amount of traditional meat products
  Interventions: Other: Traditional meat products

INTERVENTIONS:
Other: Functional meat products
  Arms: Functional meat products with healthy lipids from olive oil
Other: Traditional meat products
  Arms: Traditional meat products

SUMMARY:
Nutritional clinical trial to evaluate the effectiveness of different functional meat products on the nutritional status of healthy people

DETAILED DESCRIPTION:
Different studies have revealed that many chronic pathologies including cardiovascular disease, diabetes, autoimmune disorders, cancer, obesity or neurological diseases, could be influenced by different dietary components, such as lipids. Thus, looking for ways to substitute healthier lipids for fats that contain high amounts of cholesterol, saturated fatty acids or trans fat, could be of great interest in the prevention of chronic diseases.

Currently, meat and meat products, especially those where the fat is one of the main ingredients of the formulation, are perceived as unhealthy foods associated with increased risk of cardiovascular disease, cancer and obesity development. This is mainly due to their content of fat, trans fat, high percentage of saturated fatty acids, and cholesterol. Examples include sausages, meat spreads, salami or mortadella. Interestingly, despite the negative perception, meat and meat products continue to hold a relevant position in the diet of the developed countries. Indeed, the group "meat, poultry, deli meats and offal" contribute to the 17% of the total dietary fat intake of the Spanish population. Moreover, the consumption of deli meats and other meat products represents 5.8% of the total caloric intake. These values support the increased interest in evaluating the effect of improving the composition of these products in the prevention of disease.

Overweight and obesity are main public health concerns worldwide. They both contribute to the development of numerous diseases increasing the morbidity and mortality rates of the adult population. In this context, it is suggested that the incorporation of healthier fats may be of great interest in the prevention of these conditions. Thus, usage of lipids from olive oil as fats replacements in meat products could be an interesting strategy for the prevention and treatment of overweight and obesity.

A randomized, controlled, nutritional intervention is proposed to evaluate the effect of functional meat products on body composition and lipid profile in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 - 65 years old.
* BMI >20<27
* Adequate education level and comprehension of the clinical study.
* Willingness to participate in the study as a volunteer and to provide written consent.

Exclusion Criteria:

* Diagnosis of Type I Diabetes .
* BMI >27
* Dyslipidemia under pharmacological treatment.
* High blood pressure.
* Dementia, neurological disease or reduction of cognitive function.
* Severe illness (hepatic disease, renal disease, etc.).
* Refusal to consume the experimental or control meat products (e.g. Vegetarians)
* Refusal to follow healthy eating guidelines.
* Taking medications that could affect the lipid and glycemic profiles (statins, fibrate, diuretics, corticoids, anti-inflammatory, hypoglucemic or insulin) 30 days before the beginning of the study.
* Taking medications or substances for weight loss management (15 days before the beginning of the study).
* Consideration to follow a weight loss diet during the duration of the study.
* Pregnancy or lactation.
* High intake of alcohol.
* Any other exclusion criteria that the main investigator considers relevant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in waist circumference | Before and after 8 weeks
  The waist circumference (WC) was measured using a Seca 201 inelastic tape (Quirumed, Valencia, Spain).

SECONDARY OUTCOMES:
Changes in lipid profile | Before and after 8 weeks
  To evaluate lipid improvements the following measurements will be taking into account:
  * Triglycerides
  * Total Cholesterol
  * Low Density Lipoprotein
  * Very Low Density Lipoprotein
  * High Density Lipoprotein
  * Apolipoprotein B100 Apolipoprotein E
  * Free fatty acids
Changes in fat depots | Before and after 8 weeks
  To evaluate changes in fat depots leptin levels will be measured
Changes in blood clotting and endothelial function | Before and after 8 weeks
  To evaluate changes in blood clotting and endothelial function will be taken into account:
  * PAI I
  * Fibrinogen
Product safety | Before and after 8 weeks
  To con trol the safety of the products the following variables will be measured:
  * Urea
  * Creatinine
  * GOT
  * GPT

CONTACTS AND LOCATIONS:
Locations (1):
- IMDEA-Food, Madrid, Madrid, Spain

REFERENCES:
- [Background] Nagao T, Watanabe H, Goto N, Onizawa K, Taguchi H, Matsuo N, Yasukawa T, Tsushima R, Shimasaki H, Itakura H. Dietary diacylglycerol suppresses accumulation of body fat compared to triacylglycerol in men in a double-blind controlled trial. J Nutr. 2000 Apr;130(4):792-7. doi: 10.1093/jn/130.4.792. PMID 10736331
- [Background] Pearson AM. (1997). Principles and applications in production of reduced and low fat products. In: Production and processing of healthy meat, poultry and fish products. Advances in meat research. Vol 11. Pearson AM, Dutson TR (Eds). Blackie Academic & Professional
- [Background] Rudkowska I, Roynette CE, Demonty I, Vanstone CA, Jew S, Jones PJ. Diacylglycerol: efficacy and mechanism of action of an anti-obesity agent. Obes Res. 2005 Nov;13(11):1864-76. doi: 10.1038/oby.2005.229. PMID 16339116
- [Background] Saito S, Yamaguchi T, Shoji K, Hibi M, Sugita T, Takase H. Effect of low concentration of diacylglycerol on mildly postprandial hypertriglyceridemia. Atherosclerosis. 2010 Dec;213(2):539-44. doi: 10.1016/j.atherosclerosis.2010.07.062. Epub 2010 Aug 19. PMID 20837352